CLINICAL TRIAL: NCT06623994
Title: Bridging the Treatment Gap by Expanding Access to Care for People With Epilepsy in Kenya (BEACON)
Acronym: BEACON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jane von Gaudecker, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23924
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2025-08-18 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care Group (No Intervention): The current standard of care will be delivered. Care will be provided to the individual at the health facility by a clinician (clinical officer in levels 3, 4 & 5, medical officer in level 5), including regular consultation, vital signs, clinical history, physical examination, and prescriptions as required to control seizures.
- BEACON Group (Experimental): Those randomized to the BEACON group will receive care from clinicians who received training in epilepsy management and care. Epilepsy management tasks will be shared among the trained clinicians (e.g., nurses will offer care at all levels). ASMs used will be the same as usual care. Details about the patient will be entered in the medical records system to help with return appointment patient tracking and follow-up. Two days before the follow-up appointment date, participants will be contacted via phone or text messaging to remind them about the follow-up appointments. If participants cannot be contacted via phone a day before the appointment, the local CHW will make attempts to contact them at home. Participants who miss the appointment will be contacted again, and another appointment date will be given.
  Interventions: Behavioral: Task sharing with Epilepsy Medical Record Systems

INTERVENTIONS:
Behavioral: Task sharing with Epilepsy Medical Record Systems — Training multiple cadres of healthcare workers in epilepsy treatment and management to enable a team-based approach to address access to care. Task sharing will be supported by epilepsy medical records system with patient tracking data to support care retention
  Arms: BEACON Group

SUMMARY:
This cluster randomized trial aims to learn about the effectiveness of task-sharing supported by an epilepsy medical records system (EMRS) (hereafter referred to as BEACON) with patient-tracking data in improving treatment adherence and retention in care in people with epilepsy in western Kenya.

DETAILED DESCRIPTION:
Epilepsy is a serious neurological condition and a major cause of morbidity and mortality. Globally, epilepsy prevalence is highest in sub-Saharan Africa, and Kenya has a high disease burden. Delay in treatment initiation and non-adherence increase disease-related burden in terms of low quality of life, high healthcare costs, risk for seizure-related injuries, and premature death

The BEACON intervention is grounded in existing evidence-based intervention. Task-sharing, an intervention advocated by the World Health Organization and the Institute of Medicine. Researchers will compare patients receiving the BEACON intervention to those receiving usual care to see if there are any differences in treatment adherence and retention in care between the groups. Researchers will test BEACON's ability to: (1) improve care retention and treatment adherence; and (2) reduce seizure severity and perceived stigma and improve quality of life (QoL). The cost-effectiveness of the intervention will also be assessed. Data will be collected at baseline, 12 and 18 months (if warranted).

This project will also build clinical and research capacity for epilepsy work in western Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥12 years
* Residents of Busia or Trans Nzoia County
* Diagnosed with possible epilepsy through initial screening and confirmed diagnosis by an epilepsy-trained professional with the BEACON project or physician
* Have a diagnosis of epilepsy but are not adherent to antiseizure medication treatment.

Exclusion Criteria:

* Individuals receiving care from a neurosurgeon or neurologist for a serious brain disorder
* Unable or unwilling to provide voluntary informed consent or assent (12-18 years)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 530 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
VOILS: Domains of Subjective Extent of Nonadherence (DOSE-Nonadherence) | Baseline; 1 year; upto 18-months-if warranted
  Changes in self-reported adherence to antiseizure medication at one year from baseline as assessed using a two-domain self-report measure of medication non-adherence tool
Antiseizure medication blood levels | Baseline; 1 year; upto 18-months-if warranted
  Blood concentration of antiseizure medications will be measured as a direct method of assessing medication adherence. A blood sample (2ml) will be collected to measure adherence.
Number of participants retained in care | 1 year; upto 18-months-if warranted
  For the BEACON group, an electronic medical record system will be used to track follow-up status, patient reminders and retention in care. For usual care, participant follow-up status will be recorded in the patient chart to mimic real-world practice.
  Retention in care status will be recorded as yes/no. Retention in care will be defined as at least 1 follow-up visit 6 months -1 year after first visit

SECONDARY OUTCOMES:
Liverpool Seizure Severity Scale 2.0 | Baseline; 1 year; upto 18-months-if warranted
  NINDS Common Data Elements tool to measure perception of seizure severity. The 12-item tool measures the number of seizures and how the patient rates its severity. The tool also measures the nature of their seizures and the effects of their seizures.
  Total score is the sum of individual item scores, with higher scores indicating more severe or impactful seizures. The total score ranges from 0 (no seizures) to 100 (most severe possible)
World Health Organization Quality of Life (WHOQOL-BREF) | Baseline; 1 year; upto 18-months-if warranted
  The 26-item scale measures four domains related to quality of life: physical health, psychological, social relationships, and environment. The responses for each item are on a 5-point Likert scale. The raw scores are then transformed to a 0 to 100 scale for easier interpretation, with higher scores indicating better quality of life in that domain.
Kilifi Epilepsy Perceived Stigma Scale (KESS) | Baseline; 1 year; upto 18-months-if warranted
  This 15-item scale which was developed in Kenyan setting, measures perceived stigma. Specifically, the tool assesses (1) not relating well with family members, 2) not being accepted by peers) and 3) not being taken seriously by other people. Each item is scored on a 3-point Likert scale, leading to a total possible score ranging from 0 to 30. Higher the score greater the perceived stigma.
European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) | Baseline, one month, 6 months, 1 year, 18 months (if warranted)
  The EQ-5D-3L tool will be used to estimate the impact of BEACON in terms of costs per quality-of-life years gained relative to usual care. The scale ranges from 0 to 100 with 100 being the best health.

OTHER OUTCOMES:
Seizure-safety checklist | Each visit
  Using a 5-item questionnaire, participants will be assessed for any seizure-related injury, including type of injury and duration.
Mortality | 1 year
  Death by the end of 1-year follow-up. It will be reported as Alive: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Jane von Gaudecker, PhD, Principal Investigator — Indiana University
Locations (1):
- Moi University, Eldoret, Kenya